CLINICAL TRIAL: NCT02417948
Title: Improving Sun-Protective Behaviors and Skin Self-Examinations Among African Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CASE1615; NCI-2015-00481 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CASE1615 (Other: Case Comprehensive Cancer Center); P30CA043703 (NIH)
Record Dates: First submitted 2015-04-13; First posted 2015-04-16 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Skin Carcinoma; Skin Melanoma
MeSH Terms: conditions — Melanoma | interventions — Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (educational brochure, online educational tutorial) (Experimental): Participants receive a skin cancer educational and preventive brochure distributed by the National Cancer Institute and watch a 30-minute online tutorial video called X-Plain about skin cancer, preventative behaviors, and skin self-examinations.
  Interventions: Other: Written Educational Brochure; Other: Online educational video
- Arm II (educational brochure) (Active Comparator): Participants receive an educational brochure as in Arm I.
  Interventions: Other: Written Educational Brochure

INTERVENTIONS:
Other: Written Educational Brochure — Receive brochure with skin cancer education and preventative information
  Other Names: Education for Intervention; Intervention, Educational
Other: Online educational video — Watch 30-minute online tutorial video about skin cancer, preventive behaviors, and skin self-examinations
  Other Names: video intervention; X-Plain
  Arms: Arm I (educational brochure, online educational tutorial)

SUMMARY:
This randomized clinical trial uses an educational brochure and online tutorial program to assess sun-protective behavior and skin self-examination among African Americans. Skin cancer is very common among African Americans, with a disproportionately high mortality rate. Providing a brochure and an online educational program about sun-protective behaviors may encourage African Americans to take preventative measures against skin cancer, help improve early skin cancer detection, determine how far the disease has spread, and plan the best treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess whether an educational brochure and online program will increase sun-protective behaviors among African-American patients who present at the general dermatology clinic.

SECONDARY OBJECTIVES:

I. To assess whether the educational brochure and online program will improve skills for skin self-examinations among African-American patients who present at the general dermatology clinic.

OUTLINE: Participants are assigned to 1 of 2 arms.

ARM I: Participants receive a skin cancer educational and preventive brochure distributed by the National Cancer Institute and watch a 30-minute online tutorial video called X-Plain about skin cancer, preventative behaviors, and skin self-examinations.

ARM II: Participants receive an educational brochure as in Arm I.

After completion of study, participants are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Self-identified African-Americans who are literate and fluent in English

Exclusion Criteria:

* Non-African-Americans
* English illiteracy
* non-fluency in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2015-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change in sunscreen use among African-American patients | Baseline to day 30
  Change in sun-protective behaviors among African-American patients. Measured by sunscreen use. All responses for questions about sun-protective behaviors are on a 5-point Likert scale. Summary scores will be created at baseline and short-term (1 month) follow-up for both control and treatment groups. The outcome variable is a continuous variable. Treatment scores individuals on the intervention group will be compared. T-tests will be used to compare mean scores for sun-protective behaviors between control and treatment groups.
Change in apparel use when exposed to sun among African-American patients | Baseline to day 30
  Change in sun-protective behaviors among African-American patients. Measured by apparel use when exposed to sun. All responses for questions about sun-protective behaviors are on a 5-point Likert scale. Summary scores will be created at baseline and short-term (1 month) follow-up for both control and treatment groups. The outcome variable is a continuous variable. Treatment scores individuals on the intervention group will be compared. T-tests will be used to compare mean scores for sun-protective behaviors between control and treatment groups.
Change in frequency of tanning among African-American patients | Baseline to day 30
  Change in sun-protective behaviors among African-American patients. Measured by frequency of tanning. All responses for questions about sun-protective behaviors are on a 5-point Likert scale. Summary scores will be created at baseline and short-term (1 month) follow-up for both control and treatment groups. The outcome variable is a continuous variable. Treatment scores individuals on the intervention group will be compared. T-tests will be used to compare mean scores for sun-protective behaviors between control and treatment groups.

SECONDARY OUTCOMES:
Change in skin self-examinations among African-American patients as measured by knowledge, behavior and anxiety | Baseline to day 30
  Analyzed by looking at increase or decrease in skin self-examinations the patients report from pre-intervention to post-intervention. Performance of skin self-examination is measured by knowledge, behavior, and anxiety. Most responses for questions about skin self-examinations are on a 5-point Likert scale, while some are yes/no or true/false. Summary scores will be created at baseline and short-term (1 month) follow-up for both control and treatment groups. The outcome variable is a continuous variable. T-tests will be used to compare mean scores for skin self-examinations between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Bordeaux, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Case Comprehensive Cancer Center, Cleveland, Ohio, United States